CLINICAL TRIAL: NCT00753064
Title: Comparative Study of Efficacy of Antiscorpion Venom Serum(AScVS)vs Prazosin in the Management of Severe Scorpion(Mesobuthus Tamulus Concanesis Pocock)Envenomation and Evaluation of Effects of the Combination of AScVS + Prazosin Therapy.
Brief Title: AScVS and/ or Prazosin for Scorpion Envenomation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haffkine Bio-Pharmaceutical Corporation Ltd. (Industry)
Responsible Party: Dr. Vivek Shridhar Natu., Vijayshree hospital, Umroli, Chiplun, Ratnagiri, Maharashtra, India. 415702.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AScVS vs Prazosin
Record Dates: First submitted 2008-09-14; First posted 2008-09-16 (Estimated); Last update posted 2008-09-16 (Estimated); Status verified 2008-09

CONDITIONS: Scorpion Envenomation
Keywords: Red Scorpion envenomation; Composite clinical scoring system; AScVS; Prazosin; Superiority
MeSH Terms: conditions — Scorpion Stings | interventions — Prazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- AScVS (Active Comparator): a clinical scoring system for dose requirement for AScVS is evolved based on sweating, pulse rate, respiratory rate, blood pressure, CNS effects and presence of priapism. Computed doses were given according to clinical grading as intravenous bolus slowly.
  Interventions: Drug: Antiscorpion venom serum(AScVS).
- Prazosin. (Active Comparator): Prazosin therapy Prazosin (30 micrograms/Kg/dose): 500 micrograms for pediatric patient, and 1mg for adult patients) will be given every 3 hourly orally till complete recovery.
  Interventions: Drug: T.Prazosin
- AScVS + Prazosin (Active Comparator): Combination AScVS and Prazosin therapy In this group, AScVS therapy will be given as mentioned in AScVS therapy group and in addition, prazosin (500 micrograms for pediatric patient and 1mg for adult patients,30 micrograms/Kg/dose) every 3 hourly will be given.
  Interventions: Drug: AScVS + Prazosin

INTERVENTIONS:
Drug: Antiscorpion venom serum(AScVS). — AScVS therapy group
  If the score is 5 and if the patient belongs to pediatric group(>12-14): 1 vial AScVS as i.v. slow bolus after test dose If the score is 5 and if the patient is adult: 2 vials of AScVS as i.v. slow bolus after test dose. For injection, 1 vial will be dissolved in 10 ml distilled water and given over a period of 4 to 5 minutes.
  According to the scores 1 vial for pediatric and 2 vials for adult patient will be increased as shown below:
  Vials of AScVS Composite score Child Adult 5-10 2 4 > 10-15 3 6 >15- 21 4 8
  Other Names: AScVS(Haffkine)
  Arms: AScVS
Drug: T.Prazosin — Prazosin therapy Prazosin (30 micrograms/Kg/dose): 500 micrograms for pediatric patient, and 1mg for adult patients) will be given every 3 hourly orally till complete recovery.
  Other Names: T.Prazosin (sun pharma)
  Arms: Prazosin.
Drug: AScVS + Prazosin — Combination AScVS and Prazosin therapy In this group, AScVS therapy will be given as mentioned in AScVS therapy group and in addition, prazosin(500 micrograms for pediatric patient and 1mg for adult patients,30 micrograms/Kg/dose) every 3 hourly will be given.
  Other Names: AScVS (Haffkine); T. Prazosin (sun pharma)
  Arms: AScVS + Prazosin

SUMMARY:
The data available for the efficacy of AScVS and prazosin is generated through different trials done in different clinical setting. Hence it was felt worthwhile to confirm the documented efficacy of AScVS and prazosin in terms of time taken for clinical recovery in a clinical trial. Along with this, effects of both the therapies on various biochemical parameters will be recorded and compared with. It was also felt necessary to study the effect of combination on the clinical outcome.

DETAILED DESCRIPTION:
Red Scorpion (Mesobuthus Tamulus Concanesis Pocock) sting is a common medical emergency in the coastal regions of India and is a cause for considerable morbidity and mortality.

Signs and symptoms show either cholinergic or adrenergic predominance. Cholinergic symptoms are profuse sweating, priapism, bradycardia, increased salivary and bronchial secretions and vomiting. Adrenergic symptoms are transient hypertension followed by hypotension, tachycardia, tachypnoea, pulmonary edema and circulatory failure in later stages. Scorpion venom blocks voltage dependent inactivation of sodium channels, resulting in intense persistent voltage depolarization of autonomic nerves with massive release of catecholamines from adrenal medulla and parasympathetic and sympathetic nerve endings.

Prazosin a selective alpha-1 blocker is used as the treatment for scorpion sting, which can only counteract the manifestations of sympathetic over-activity. Experimentally and clinically it is seen that scorpion venom stays in the body for 24-36 hours, as Prazosin does not neutralize the venom, 3 hourly round the clock doses of prazosin and continuous I.C.U. monitoring is necessary with alpha blocker therapy. However, ideal treatment modality remains neutralization of venom in the systemic circulation.

Since 1997 enzyme refined AScVS ( Monovalent Anti-scorpion venom serum against Mesobuthus tamulus concanesis Pocock.) has been made available by Haffkine Biopharmaceuticals, Mumbai for field use. Throughout the konkan(western coastal Maharashtra, India) area the same species of scorpions responsible for fatal envenomation is found.

From 1997-2002, 48 patients of serious scorpion envenomation were treated with AScVS(1). Based on this experience a clinical scoring system for dose requirement was evolved based on sweating, pulse rate, respiratory rate, blood pressure, CNS effects and presence of priapism. In our experience computed doses given as intravenous bolus are more effective and successfully ameliorated signs and symptoms in all patients. Subsequently 16 patients were given treatment with either AScVS (n=8), Prazosin (n=5) and a combination of both (n=3) so as to compare the effects of these available treatment modalities. It was found that the patients receiving either AScVs or a combination showed a complete recovery approximately within 4 hours of onset of therapy as against patients receiving Prazosin, who required 16 hours for recovery. There was no mortality in any of the group. There was not a single incidence of anaphylaxis after administration of AScVS. Release of adrenaline in the systemic circulation by scorpion sting itself appears to be protective against the danger of anaphylaxis. The label on the AScVS vials states that the maximum dose is 3 vials, which can be given either intramuscular or by intravenous route. However we used AScVS as slow bolus intravenously and dose was decided clinically depending upon the severity of the patient condition. (maximum 10-15vials.) Based on this experience, an open labeled, randomized controlled parallel group clinical trial has been initiated. Eighty-three patients have been recruited so far, 28 patients each, in AScVS and AScVS + prazosin group and 27 patients in Prazosin group, two patients out of 27 in Prazosin group were withdrawn as both the pediatric patients (around 12 years old) developed pulmonary edema after few hours, so AScVS had to be given. The onset of relief (based on composite score) with AScVS or combination of AScVS with prazosin was early and complete recovery occurred at 4.14+/- 1.6 hrs. and 3.46+/- 1.10hours. However, in patients receiving only prazosin, the clinical score was found to worsen initially, followed by a gradual improvement and subsequent complete recovery, at 19.28 +/- 5.03 hrs. (p<0.001 vs AScVS). Recovery time with AScVS is much shorter because after complete neutralization of venom, fresh secretion of catecholamines stop and adrenaline and nor-adrenaline which are already in circulation have action as short as 1 to 2 minutes. These findings appear consistent with our clinical experience and indicate that in the near future AScVS would evolve as a safe, efficacious and life saving treatment modality for patients with severe scorpion envenomation. Use of clinical scoring system can enable the clinician to select the optimum dose of AScVS to be administered.

Neutralization of venom is thus proved to be better than therapy for complications, akin to the dictum 'prevention is better than cure'.

References:

1. Natu VS, Murthy RKK, Deodhar KP. Efficacy of species specific Antiscorpion venom serum (AScVS) against severe, serious scorpion stings (mesobuthus tamulus concanesis pocock.)-An experience from rural hospital in western Maharashtra. JAPI, 2006; 54: 283-7.

ELIGIBILITY:
Inclusion Criteria: (All of the following)

1. Patients of both sexes, in the age range of 12-65 years
2. reporting to the PHC/ hospital within 48 hours of scorpion sting and
3. associated with s/s of scorpion envenomation having composite score between 5 and 21 (as computed based on the criteria below:)

Criteria Grade Symptoms

Sweating 0 Limited to the extremity of the sting site.

1. Minimal sweating all over the body, slight nasal secretions
2. Generalized sweating with rigors and cold extremities.
3. Gen.profuse sweating,wetting of clothes and cold clammy skin.

Pulse rate 0 70- 90

1. 91 - 100
2. 101 - 120 or < 70
3. 121 - 140 or < 60 or irreg pulse
4. 141 - 160
5. > 160

Respiratory rate 0 < 20

1. 20 - 30
2. 31 - 40 without crepitations
3. 31 - 40 with crepitations
4. > 40 with crepitations
5. > 40 with crepitations and cyanosis

Blood pressure 0 120/80

1. Systolic: 121 -140 and diastolic: 81 -90
2. Systolic: 141 -160 and diastolic: 91-100
3. Syst: 161 -180 and diast: 101-110 Or syst <100
4. Syst: 181 -200 and diast: 111-120 Or syst <100
5. Syst: > 200 and diast: >120 Or syst < 60

CNS effects 0 No sensory involvement

1. Minimal tingling numbness around mouth
2. Tingling, numbness around mouth and giddiness
3. Altered sensorium, patient roudy
4. Patient semiconscious
5. Patient unconscious

Priapism 2 Slight erection 3 Strong erection

To obtain a composite score, grades for individual criterion will be added. Maximum score: 25 and minimum score: 0

Exclusion Criteria: (Any of the following)

1. Composite score less than 5 and greater than 21.
2. Grade of 5 in any of the criterion
3. Severe Pulmonary edema with oxygen saturation below 80%.
4. Severe scorpion envenomation with reporting time more than 2 days
5. Any other serious medical disease which/treatment of which may confound the results e.g. cardiac diseases, diabetes, renal diseases etc.
6. Severe anaphylactic reaction to any of the study drugs
7. Patient (or relative in case of child) not willing to participate

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Superiority of AScVS and AScVS+Prazosin was confirmed over use of Prazosin alone. | 1year 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Vivek S Natu, M.S., Principal Investigator — Vijayshree Hospital, Umroli, Chiplun, Ratnagiri, Maharashtra, India.; Dr. Santosh Kamerkar, M.S, Study Chair — Cottage Hospital Mangaon,Raigad,Maharashtra, India; Dr. Geeta Kadam, M.B.B.S., Study Chair — Cottage Hospital Mangaon,Raigad,Maharashtra, India; Dr. Vidya Kamble, M.B.B.S., Study Chair — Cottage Hospital Mangaon,Raigad,Maharashtra, India; Dr. Vikas Natu, MBBS DCH, Study Chair — Natu Hospital Chiplun,Ratnagiri, Maharashtra,India; Dr. Sanjeev Sane, MBBS DCH, Study Chair — Sane Hospital Chiplun,Ratnagiri, Maharashtra,India; Dr. Rajesh Kushte, MBBSDCH, Study Chair — Kushte Hospital Chiplun,Ratnagiri, Maharashtra,India; Dr. Sunil Thatte, M.D., Study Chair — Attending physician at Natu, Sane & Kushte Hospital Chiplun,Ratnagiri, Maharashtra,India; Dr. Uchil Dinesh, Ph.D., Study Chair — A.R.C. K.E.M. Hospital Mumbai,Maharashtra,India; Dr. Nirmala Rege, M.D., Study Chair — A.R.C. K.E.M. Hospital Mumbai,Maharashtra,India; Dr. Ravindra Bapat, M.S., Study Director — K.E.M. Hospital Mumbai,Maharashtra,India
Locations (5):
- India (5):
  - Kushte Hospital, Chiplūn, Maharashtra
  - Natu Hospital, Chiplūn, Maharashtra
  - Sane Hospital, Chiplūn, Maharashtra
  - Mangaon cottage hospital, Mangaon., Dist. Raigad., Maharashtra
  - Vijayshree Hospital,At & Po.Umroli,Tal. Chiplun., Dist. Ratnagiri., Maharashtra